CLINICAL TRIAL: NCT07096518
Title: The Effect of an Education Supported by ChatGPT Integration on Nursing Students' Knowledge and Motivation Levels Regarding Aspiration Practice
Brief Title: Effect of ChatGPT-Supported Education on Nursing Students' Aspiration Practice Knowledge and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Emine SEZGÜNSAY, Assistant Professor, Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IEU-SBF-01
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Endotracheal Aspiration; Nursing Education; Artificial Intelegence; Knowledge; Motivation
Keywords: nursing education; knowledge; endotraceal suctioning; Knowledge Retention; artificial intelligent; motivation; ChatGPT

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group, which received a ChatGPT-integrated lecture, or the control group, which received a traditional lecture. Both groups were assessed before and after the intervention. Students' motivation levels and feedback were collected immediately after the lectures, and knowledge retention was evaluated with a follow-up test conducted six weeks later. This parallel-assignment design allowed for a direct comparison between the two teaching methods.
Masking Description: Participants were not formally informed of their group assignment, but due to the nature of the intervention, masking was not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Lecture Group (No Intervention): This group received a traditional lecture based on a passive learning model, where the student is a passive recipient and the instructor is the information provider. The lecture included PowerPoint presentations, question-and-answer sessions, and video demonstrations.
- ChatGPT-Integrated Lecture Group (Experimental): This group received a structured and interactive educational lecture integrated with ChatGPT, an AI language model, enabling students to learn collaboratively through guided activities related to endotracheal suctioning. Students compared the information obtained from ChatGPT with evidence-based, up-to-date clinical guidelines and discussed the comparison results together in the classroom. The instructor provided guidance throughout the process.
  Interventions: Other: ChatGPT-Integrated Lecture

INTERVENTIONS:
Other: ChatGPT-Integrated Lecture — This group received a structured and interactive educational lecture integrated with ChatGPT, an AI language model, enabling students to learn collaboratively through guided activities related to endotracheal suctioning. Students compared the information obtained from ChatGPT with evidence-based, up-to-date clinical guidelines and discussed the comparison results together in the classroom. The instructor provided guidance throughout the process.
  Arms: ChatGPT-Integrated Lecture Group

SUMMARY:
This study was designed to examine the effects of a Chat Generative Pre-trained Transformer (ChatGPT)-integrated lecture on nursing students' knowledge, motivation, and knowledge retention related to endotracheal suctioning. The effects of this Artificial Intelligence (AI)-supported lecture were compared with those of a traditional lecture. ChatGPT, an AI-based language model, was used to provide interactive and personalized support during the learning process.

DETAILED DESCRIPTION:
This study was designed to investigate the effects of ChatGPT-integrated education on nursing students' knowledge, motivation, and knowledge retention related to endotracheal suctioning practice. Additionally, the study aimed to compare this innovative approach with traditional teaching methods and to explore students' feelings and perceptions regarding both learning experiences.

Endotracheal suctioning is a critical nursing procedure, especially in intensive care settings, to maintain airway patency and ensure adequate oxygenation. However, existing literature indicates that nursing students often find this procedure challenging and anxiety-inducing, with generally low levels of knowledge.

AI tools like ChatGPT have been reported to enhance individualized learning, critical thinking, and problem-solving skills. Therefore, integrating ChatGPT into nursing education was considered to have the potential to improve theoretical knowledge acquisition and increase students' motivation toward the lecture.

The study was conducted with third- and fourth-year nursing students enrolled in the undergraduate program at Izmir University of Economics, using a randomized controlled, quasi-experimental design. Knowledge, motivation levels, and knowledge retention were compared between control and intervention groups to evaluate the effect of ChatGPT-integrated education. Additionally, students' feedback regarding the educational experience was collected and analyzed.

Data collection instruments included the Student Information Form, the Suctioning Knowledge Questionnaire, the ARCS (Attention, Relevance, Confidence, and Satisfaction) Motivation Learning Scale, and the Student Feedback Form.

Lectures were planned separately for the control and intervention groups. The control group received traditional instruction methods such as presentations, video demonstrations, and discussions. In contrast, the intervention group accessed information and performed critical evaluations using ChatGPT. In a classroom setting, students discussed the information obtained via ChatGPT by comparing it with the latest published clinical guidelines on suctioning practice. Knowledge tests were administered before and after the lectures in both groups, and a follow-up knowledge test was conducted six weeks later to assess knowledge retention.

Data analysis was performed using SPSS version 21. Frequency analysis was conducted for categorical data, descriptive statistics for numerical data, and parametric or non-parametric tests were applied for group comparisons. The level of significance was set at 0.05. The findings aimed to evaluate the effectiveness of the educational programs and demonstrate the impact of innovative teaching approaches.

Ethical approval was obtained from the Ethics Committee for Health Sciences Research at Izmir University of Economics and the Dean's Office of the Faculty of Health Sciences. Participants were informed about the study, data confidentiality, and their right to withdraw at any time. All participants provided written informed consent. Necessary permissions were obtained for the use of validated measurement tools, and all course materials were shared with participants via the Blackboard platform.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students who are enrolled in the Surgical Units Nursing II course
* Students who voluntarily agree to participate in the study

Exclusion Criteria:

* Students who do not attend the planned lecture session
* Students who do not respond to the pre- or post-intervention surveys

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Endotracheal Aspiration Knowledge Score | Baseline (Pre-intervention) and immediately after the final session
  Participants' knowledge regarding endotracheal suctioning will be assessed before and after the educational intervention using a validated multiple-choice questionnaire. The change in knowledge scores will be used to evaluate the effectiveness of the ChatGPT-integrated structured learning model compared to the traditional lecture approach.

SECONDARY OUTCOMES:
Change in Student Motivation Level | Immediately after the educational session
  Participants' motivation related to the instructional materials will be measured immediately after the educational intervention using a validated scale. This assessment will allow comparison of learners' motivation levels in relation to instructional materials between the ChatGPT-integrated lecture group and the traditional lecture group.
Retention of Endotracheal Suctioning Knowledge at 6 Weeks | 6 weeks after the educational session
  Participants' knowledge retention regarding endotracheal suctioning will be assessed six weeks after the educational intervention using the same validated multiple-choice questionnaire. The scores will be compared between the ChatGPT-integrated lecture group and the traditional lecture group to evaluate the long-term effectiveness of the intervention.

OTHER OUTCOMES:
Qualitative Feedback from Students on Educational Experience | Immediately after the educational session
  Open-ended feedback from participants collected immediately after the educational intervention. Responses will be analyzed thematically to explore students' perceptions, experiences, and suggestions regarding the ChatGPT-integrated lecture and traditional lecture methods.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Sezgünsay, PhD, Principal Investigator — İzmir University of Economics, Department of Nursing
Locations (1):
- İzmir University of ;Economics, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional data protection policies and the educational nature of the study. Participants were not informed or consented for public data sharing.

REFERENCES:
- [Background] Shorey S, Mattar C, Pereira TL, Choolani M. A scoping review of ChatGPT's role in healthcare education and research. Nurse Educ Today. 2024 Apr;135:106121. doi: 10.1016/j.nedt.2024.106121. Epub 2024 Feb 6. PMID 38340639
- [Background] Gunawan J, Aungsuroch Y, Montayre J. ChatGPT integration within nursing education and its implications for nursing students: A systematic review and text network analysis. Nurse Educ Today. 2024 Oct;141:106323. doi: 10.1016/j.nedt.2024.106323. Epub 2024 Jul 26. PMID 39068726